CLINICAL TRIAL: NCT05498532
Title: Functional MRI Usage for Pyelo-ureteral Junction Syndrome : Results of Nancy Children Hospital Cohort
Brief Title: Functional MRI Evaluation in Pyeloureteral Junction Syndrome in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Charles Mazeaud, Praticien hospitalier universitaire, Central Hospital, Nancy, France
Other Study IDs: 2022PI108
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Stricture of Pelviureteric Juncture
Keywords: PUJS; MRI; Scintigraphy; Polar Vessel
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PUJS patients: Patients between 0 and 17 years old treated or followed for pyelo-ureteral junction syndrome.
  Interventions: Diagnostic Test: Functional MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — Anatomical MRI : T2 fiesta, SSFE, HASTE ; 3D T2 ; T1 FAT SAT ; LAVA Functional MRI : T1 FAT SAT with gadolinium
  Other Names: Renal Scintigraphy

SUMMARY:
Pyelo-ureteral junction syndrome is the most common urological abnormality in children.

Functional MRI has been evaluated several times, and had shown good correlation with scintigraphy, but tends to over estimate results. Moreover, those studies included a small number of cases. Its sensitivity to detect crossing polar vessel is limited.

We aimed to evaluate, in patients between 0 and 1 year old, the correlation between MRI and scintigraphy differential renal function.

Our secondary objectives are : evaluation of MRI performances to detect polar vessel ; comparison of surgery times depending of MRI only realisation or MRI and scintigraphy realisation.

ELIGIBILITY:
Inclusion Criteria:

* children between 0 and 17 years old
* followed for pyelo-ureteral junction syndrome

Exclusion Criteria:

* none

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 0 and 17 years old followed for pyelo-ureteral junction syndrome in the Children hospital of Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
MRI and scintigraphy differential renal function correlation | from january 2007 to december 2021
  Evaluation of differential renal function between MRI and scintigraphy in children between 0 and 1 year old ; Pearson correlation coefficient

SECONDARY OUTCOMES:
MRI and scintigraphy differential renal function correlation in operated patient | from january 2007 to december 2021
  Evaluation of differential renal function between MRI and scintigraphy in children operated for PUJS; Pearson correlation coefficient
Time difference in patient operated for PUJS depending on MRI realisation ou MRI and scintigraphy realisation | from january 2007 to december 2021
  Comparison between the mean time between MRI and surgery, and mean time between MRI, scintigraphy and surgery
performance of MRI in detecting polar vessel | from january 2007 to december 2021
  Polar vessel : comparison between MRI results and operatory observation, sensitivity et specificity analysis

CONTACTS AND LOCATIONS:
Overall Officials: Charles Mazeaud, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, Lorraine, France